CLINICAL TRIAL: NCT05661227
Title: Mechanism of Cardiac and Cerebral Function Injury in Patients With Coronary Heart Disease Caused by Intraoperative Limb Ischemia-reperfusion and Perioperative Organ Function Protection Strategy
Brief Title: Mechanism of Cardiac and Cerebral Function Injury Caused by Intraoperative Limb Ischemia-reperfusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Liuxin2022
Record Dates: First submitted 2022-11-17; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Ischemic Reperfusion Injury
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- C group (Sham Comparator): Before induction of anesthesia, general anesthesia was performed after ultrasound-guided femoral nerve block
  Interventions: Drug: 0.9% Sodium chloride
- DEX group (Experimental): Before induction of anesthesia, general anesthesia was performed after ultrasound-guided femoral nerve block. Dexmedetomidine 0.8μg/kg was pumped intravenously for 10min 15min before induction of anesthesia, and then continued to be infused at 0.5μg/ (kg·h) until 30min before the end of surgery
  Interventions: Drug: Dexmedetomidine
- ERIPC group (Experimental): Before induction of anesthesia, ultrasound-guided femoral nerve block was performed, and then general anesthesia was performed. After induction of anesthesia, orthopedic tourniquet was tied and inflated to 200 mmHg(1 mmHg=0.133 kPa) for 5 min and deflated for 5 min, and three cycles were repeated
  Interventions: Device: Tourniquet(Early)
- LRIPC group (Experimental): An orthopedic pressure tourniquet was placed on the lower extremity 24 h before surgery and inflated to 200 mmHg for 5 min and deflated for 5 min. Three cycles were repeated
  Interventions: Device: Tourniquet(Late)

INTERVENTIONS:
Drug: Dexmedetomidine — Whether apply DEX or not
  Other Names: DEX
  Arms: DEX group
Drug: 0.9% Sodium chloride — Whether apply DEX or not
  Other Names: NS
  Arms: C group
Device: Tourniquet(Early) — Timing of tourniquet application
  Arms: ERIPC group
Device: Tourniquet(Late) — Timing of tourniquet application
  Arms: LRIPC group

SUMMARY:
As a simple auxiliary tool for lower extremity orthopedic surgery, tourniquet can effectively reduce intraoperative bleeding and ensure the clarity of the operative field, effectively shorten the operation time and improve the operation efficiency. The extensive use of tourniquets in lower extremity surgery will not only cause local paralysis, pain and other complications, but also bring about postoperative complications such as large drainage volume and deep vein thrombosis. Recent studies have found that tourniquet induced ischemia-reperfusion injury not only affects the local tissue structure and function of skeletal muscle, but also causes reperfusion injury in distant organs (such as heart, lung and brain). Therefore, improving tourniquet ischemia-reperfusion injury after knee replacement is of great significance to improve the quality of life of patients during the perioperative period. Therefore, the aim of this study was to investigate the effects of dexmedetomidine and tourniquet pretreatment on myocardial injury and brain injury caused by lower extremity ischemia-reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TKA under general anesthesia
* Voluntarily sign the informed consent
* ASA Grade I to III
* BMI 18-28 kg/m2

Exclusion Criteria:

* Congenital heart disease or history of cardiac surgery, heart conduction disease, frequent ventricular/atrial premature beats, atrial fibrillation and other serious arrhythmias
* Severe liver disease and kidney disease
* Temporary and permanent pacemaker implantation
* Patients with serious central nervous system diseases or serious mental disorders
* Recent history of sedation, antidepressant or opioid use
* Body mass index >35kg/m2
* Participants in other clinical trials within 1 month prior to study enrollment.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
SOD | Baseline to day2
  Superoxide dismutase
MDA | Baseline to day2
  Malonaldehyde
IL-6 | Baseline to day2
  Interleukin- 6
TNF-α | Baseline to day2
  Tumor necrosis factor-α
hs-Tn | Baseline to day2
  High sensitive troponin
BDNF | Baseline to day2
  Brain-derived neurotrophic factor

SECONDARY OUTCOMES:
HRV | Baseline to day2
  HeartRateVariability
PRR | Baseline to day2
  Pulse Repetition Rate
BP | Baseline to day2
  Blood Pressure（both systolic and diastolic blood pressure will be measured）
SpO2 | Baseline to day2
  Peripheral capillary oxygen saturation
VAS | Baseline to day2
  Visual Analogue Scale/Score(Draw a 10cm horizontal line on the paper. One end of the horizontal line is 0, indicating no pain; the other end is 10, indicating severe pain; the middle part indicates pain. Different degrees of pain. Let the patient draw a mark on the horizontal line according to his own feelings to indicate the degree of pain.)
MMSE | Baseline to day2
  Mini-mental State Examination（The scale includes the following seven aspects: time orientation, place orientation, instant recall, attention and computational power, delayed memory, language, and whether to answer correctly or not. The test scores are closely related to the educational level. The normal threshold is more than 20 points, and the junior high school and above are more than 24 points）

CONTACTS AND LOCATIONS:
Overall Officials: PengChen Wang, Study Chair — Hebei Medical University Third Hospital
Locations (1):
- The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No